CLINICAL TRIAL: NCT06012812
Title: A Multicenter, Open-label, Extended Study Evaluating the Safety and Efficacy of SHR-1819 Injection in Adult Subjects With Moderate to Severe Atopic Dermatitis Who Have Previously Participated in SHR-1819 Studies for the Treatment of Atopic Dermatitis
Brief Title: A Study to Extend Efficacy and Safety of SHR-1819 Injection in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1819-203
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1819 injection (Experimental)
  Interventions: Drug: SHR-1819 injection

INTERVENTIONS:
Drug: SHR-1819 injection — SHR-1819 injection 300 mg Q2W

SUMMARY:
This study is a multicenter, open-label, extended study to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of SHR-1819 injection in adult subjects with moderate to severe atopic dermatitis who have previously participated in the SHR-1819 injection study for atopic dermatitis (defined as the main study, referred to as the main study hereinafter).

ELIGIBILITY:
Inclusion Criteria:

1. The age of 18~75 years old at the time of signing the informed consent form (including the values at both ends), gender is not limited；
2. Previous atopic dermatitis, (1) participation in a complete main study; or (2) subjects who prematurely terminate primary study therapy for reasons other than SHR-1819 injection are required to complete a last safety follow-up or withdrawal from the visit, and the investigator assesses that the influencing factor has been eliminated/no longer affects the participant's participation in the extended study. Participants were required to meet the main study inclusion criteria for the main study；
3. Be able to apply a topical emollient (moisturizer) continuously for at least 7 consecutive days before the first dose and continue to use it for the duration of the study;
4. Be able to sign informed consent forms, understand and agree to follow the requirements of the study and the trial process.

Exclusion Criteria:

1. Pregnant or lactating women；
2. Female subjects of childbearing potential and male subjects whose partners are women of childbearing age have a plan to donate sperm/eggs from the signing of the informed consent form until 3 months after the last dose of the trial drug, or refuse to comply with the relevant contraceptive requirements;
3. A history of alcohol abuse or illicit drug abuse within 6 months prior to screening;
4. Hypersensitivity to the study drug or any ingredient in the study drug；
5. Diagnosed within 6 months prior to screening or judged by the investigator to have a suspected immunosuppressive disease;
6. Oral or parenteral systemic antimicrobials are used within 2 weeks before the first dose；
7. Suspected or confirmed active tuberculosis (TB);
8. Have malignancy or history of malignancy prior to screening；
9. Major surgery was performed within 3 months prior to screening, or major surgery was planned during the study；
10. There are currently significant abnormal laboratory test results, severe concomitant diseases, and other circumstances that the investigator considers inappropriate to participate in this trial;
11. There were treatment-related adverse events leading to discontinuation of treatment and study drug-related SAEs in the main study, and the investigator or sponsor medical department considered that continuing to participate in extended therapy would pose an unacceptable safety risk to participants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) (per person-year) | Up to 60 weeks

SECONDARY OUTCOMES:
Serious Adverse Event (SAE) during treatment (per person-year) | Up to 60 weeks
Adverse Events of Special Interest (AESI) during treatment (per person-year) | Up to 60 weeks
Proportion of participants with a Global Assessment (IGA) score of 0 or 1 (0-4 scale) per visit | Up to 60 weeks
Time to first remission (remission defined as IGA = 1 or 0 after treatment) in this study (for participants visiting 2 baseline IGAs ≥2) | Up to 60 weeks
Proportion of participants with at least 1 remission in this study | Up to 60 weeks
Time to first relapse in this study (relapse defined as IGA = 3 or 4 points after remission) (for participants with Visit 2 baseline IGA ≥ 2) | Up to 60 weeks
The concentration of SHR-1819 in serum :Cmax | From the beginning of administration to the 60h week
Immunogenic endpoint: evaluate the incidence and timing of ADA positivity for SHR-1819 | From the beginning of administration to the 60th week

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided